CLINICAL TRIAL: NCT04681833
Title: A Randomised, Double-blind, Placebo-controlled, Dose-ranging Phase II Study in 60 to 80-Year-Old Adults to Assess the Safety and Immunogenicity of BARS13
Brief Title: Safety and Efficacy of BARS13 in the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advaccine (Suzhou) Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADVA-BARS13-002
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); BARS13; Vaccines; Virus Diseases
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of one arm, and one dose of placebo by IM injection to the deltoid region of the other arm, given sequentially (10 μg rRSV G protein/10 μg CsA in total for each vaccination) on Day 1 and 29.
  Placebo: One dose administered by IM injection to both arms, on Day 1 and 29.
  Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of each arm, given sequentially (20 μg rRSV G protein/20 μg CsA in total for each vaccination) on Day 1 and 29.
  Placebo: One dose administered by IM injection to both arms, on Day 1 and 29.
  Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of each arm, given sequentially (20 μg rRSV G protein/20 μg CsA in total for each vaccination) on Day 1, Day 29 and Day 57.
  Placebo: One dose administered by IM injection to both arms, on Day 1, Day 29 and Day 57.
Who Masked: Participant, Investigator
Masking Description: This study is double-blinded. Sealed participant-specific code break envelopes will be produced by the unblinded statistician so that the treatment assigned to each participant can be obtained if required, in an emergency only, where knowledge of the randomisation code is required to provide appropriate treatment. The code break envelopes will be retained at the clinical unit in a secure, accessible location. Those blinded to study drug assignment include the sponsor, the PI, clinical study personnel participating in participants' care or clinical evaluations, and the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1: BARS13 low repeat dose (Experimental): Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of one arm, and one dose of placebo by IM injection to the deltoid region of the other arm, given sequentially (10 μg rRSV G protein/10 μg CsA in total for each vaccination) on Day 1 and 29.
  Interventions: Drug: Recombinant Respiratory Syncytial Virus Vaccine (BARS13) /placebo
- Cohort 1: BARS13 placebo low repeat dose (Placebo Comparator): Placebo: One dose administered by IM injection to both arms, on Day 1 and 29.
  Interventions: Drug: Placebo
- Cohort 2: BARS13 high repeat dose (Experimental): Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of each arm, given sequentially (20 μg rRSV G protein/20 μg CsA in total for each vaccination) on Day 1 and 29.
  Interventions: Drug: Recombinant Respiratory Syncytial Virus Vaccine (BARS13)
- Cohort 2: BARS13 placebo high repeat dose (Placebo Comparator): Placebo: One dose administered by IM injection to both arms, on Day 1 and 29.
  Interventions: Drug: Placebo
- Cohort 3: BARS13 high repeat multiple dose (Experimental): Active: One dose of 10 μg rRSV G protein/10 μg CsA administered by IM injection to the deltoid region of each arm, given sequentially (20 μg rRSV G protein/20 μg CsA in total for each vaccination) on Day 1, Day 29 and Day 57.
  Interventions: Drug: Recombinant Respiratory Syncytial Virus Vaccine (BARS13)
- Cohort 3: BARS13 placebo high repeat multiple dose (Placebo Comparator): Placebo: One dose administered by IM injection to both arms, on Day 1, Day 29 and Day 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Respiratory Syncytial Virus Vaccine (BARS13) /placebo — Low Repeat Dose
  Arms: Cohort 1: BARS13 low repeat dose
Drug: Recombinant Respiratory Syncytial Virus Vaccine (BARS13) — High Repeat Dose/High Repeat Multiple Dose
  Arms: Cohort 2: BARS13 high repeat dose; Cohort 3: BARS13 high repeat multiple dose
Drug: Placebo — Liquid diluent/Lyophilised Powder
  Arms: Cohort 1: BARS13 placebo low repeat dose; Cohort 2: BARS13 placebo high repeat dose; Cohort 3: BARS13 placebo high repeat multiple dose

SUMMARY:
Advaccine Clinical Research are developing a vaccine called BARS13 for the active immunisation of infants (aged 6 months to 5 years old) and the elderly (aged 60-80 years old) for the seasonal prevention of Respiratory Syncytial Virus (RSV) infection. A total of 125 volunteers aged 60 - 80 years (inclusive) will be enrolled in this study, and will be divided into 3 groups (or 'cohorts') of 40 people (cohort 1 and 2) and 45 people (cohort 3). The aim of the study is to evaluate the safety and tolerability of BARS13 in this age group.

DETAILED DESCRIPTION:
Advaccine Clinical Research is developing a recombinant Respiratory Syncytial Virus (rRSV) vaccine - BARS13 for the protection of the elderly from RSV infection.

This is a two centre, randomised, double-blind, placebo-controlled study in healthy adults aged 60-80 years old to evaluate the safety and immunogenicity of the rRSV investigational vaccine, BARS13.

This study will be conducted in two centres in Australia with CMAX as the coordinating site.

A total of up to 125 eligible participants will be enrolled administered by IM injection to the deltoid region of the arm. Cohort 1 (low repeat dose) includes one dose of 10micrograms of the vaccine on one arm and one dose of placebo on the other arm given sequentially on Day 1 and 29. Cohort 2 (high repeat dose) includes one dose of 10micrograms of the vaccine on each arm given sequentially on Day 1 and 29. Cohort 3 (high repeat multiple dose) includes one dose of 10microgarms of vaccine to each arm sequentially on Day 1, 29 and 57.

ELIGIBILITY:
Inclusion:

Participants who meet all of the following criteria at screening are eligible to participate in the study:

1. Healthy male or female adults, or adults with stable chronic disease aged 60 to 80 years old, inclusive. Stable disease includes adults with no new diagnosis, hospitalization or changes in medication in the preceding 3 months. Adults with stable, Stage 1 chronic obstructive pulmonary disease (COPD) are eligible for this study provided they are not using inhaled or systemic corticosteroids.
2. Body mass index (BMI) ≤40 kg/m2.
3. Screening 12-lead electrocardiogram (ECG) must be within normal range (QT interval corrected using Fridericia's formula [QTcF] males ≤ 450 msec; females ≤ 470 msec) or with abnormalities, which are not hazardous to the patient according to the opinion of the Investigator at the screening visit.
4. Hematology, serum chemistry, coagulation and urinalysis test results not deviating from the normal reference range by age and gender to a clinically relevant extent at screening.
5. Systolic blood pressure in the range of 90 to 160 mmHg (inclusive) and diastolic blood pressure in the range of 50 to 95 mmHg (inclusive) after 5 minutes in supine position at the screening visit. (May be repeated twice, if abnormal values were recorded in the first instance, at the discretion of the PI).
6. Willing and able (on both a physical and cognitive basis) to give informed consent prior to study enrolment.
7. Able to comply with study requirements, including access to transportation for study visits.
8. Access to inbound and outbound telephone communication with caregivers and study staff.
9. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent or, if engaged in sexual relations with a person of child-bearing potential, the participant and his partner must use an acceptable, highly effective, contraceptive method from screening and for a period of at least 3 months after the last dose of study drug. Acceptable methods of contraception are the use of condoms and an effective contraceptive for the female partner that could include surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception, or intrauterine contraception/device. The PI or appropriate designee is to assess the adequacy of methods of contraception on a case-by-case basis.
10. Females must be of nonchildbearing potential i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone level ≥40 IU/L at the screening visit).

Exclusion:

Participants who meet any of the following criteria are not eligible to participate in the study:

1. Participation in research involving investigational product (IP) (drug / biologic / device) within 45 days before the planned date of the Day 1 vaccination.
2. History of a serious reaction to any prior vaccination.
3. Received any vaccine other than an inactivated or live attenuated influenza vaccine or coronavirus SARS-COV-2 (COVID-19) vaccine (not in a clinical trial setting) in the 4 weeks preceding the first study vaccination; or any RSV vaccine at any time or who plan to receive any non-study vaccines within 28 days of the last dose of study vaccine. Influenza vaccine and coronavirus SARS-COV-2 (COVID-19) vaccine should not be given within 14 days of each dose of study vaccine.
4. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
5. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical and nasal glucocorticoids will be permitted.
6. Positive testing for active HIV, HBsAg, HCV, Quantiferon (TB infection).
7. Positive urine drug screen at screening, or pre-vaccination for any drug of abuse unless there is an explanation acceptable to the PI (e.g., the participant stated in advance that they consumed a prescription or over the counter product which contained the detected drug) and/or the participant had a negative urine drug screen on retest by the pathology laboratory.
8. A positive alcohol breathalyzer test at screening or pre-vaccination.
9. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
10. Acute disease at the time of enrolment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥38.0°C on the planned day of vaccine administration).
11. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse (regular consumption of > 10 units of alcohol/week [men and women]; 1 unit = 237 mL of beer, 25 mL shot of 40% spirit or a 125 mL glass of wine. A standard drink contains 10 g of alcohol).
12. Birthmarks, tattoos, wound or other skin conditions over the deltoid region of either arm that, in the PI's opinion, could reasonably obscure and interfere with evaluation of local injection site reactions.
13. Subject with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren syndrome, idiopathic thrombocytopenic purpura, autoimmune glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (Type 1), Crohn's disease or ulcerative colitis.
14. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic, cognitive, or psychiatric conditions deemed likely to impair the quality of study compliance or safety reporting).
15. History of any chronic respiratory illness, including current diagnosis of asthma within 2 years, COPD ≥ Stage 2, exercise induced wheezing, reactive airway disease, emphysema, chronic bronchitis or cystic fibrosis. Asthma diagnosed > 2 years ago is allowed at PI discretion if the asthma is considered well controlled as per the Asthma Australia Control Tool (score of ≥20 out of 25). Inhaled corticosteroids are allowed provided dose is considered <10 mg prednisolone equivalent.
16. Any respiratory illness (e.g., cough, sore throat, dyspnea, wheezing or nocturnal awakenings to respiratory symptoms) within 14 days prior to receiving the first dose of study vaccination.
17. Any active pulmonary infection or other inflammatory conditions, even in the absence of febrile episodes, within 14 days prior to the first study vaccination.
18. Any other condition or prior therapy that in the opinion of the PI would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of vaccine-related AEs, including the following solicited AEs | From baseline (Day 1) to the end of Day 7.
  Incidence and severity of local reactions (pain, tenderness, erythema, swelling, other e.g., ulceration, scabs, bruising, itching and paraesthesia) at the site of vaccination; Incidence and severity of systemic reactions (fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea, diarrhea, light-headedness, dizziness, hypersensitivity and headache). Any 'solicited' AE with onset outside the specified 7-day period of follow-up will be reported as an unsolicited AE.
Incidence and severity of vaccine-related AEs, including the following solicited AEs | From Day 28 to the end of Day 35.
  Incidence and severity of local reactions (pain, tenderness, erythema, swelling, other e.g., ulceration, scabs, bruising, itching and paraesthesia) at the site of vaccination; Incidence and severity of systemic reactions (fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea, diarrhea, light-headedness, dizziness, hypersensitivity and headache). Any 'solicited' AE with onset outside the specified 7-day period of follow-up will be reported as an unsolicited AE.
Incidence and severity of vaccine-related AEs, including the following solicited AEs | From Day 57 to the end of Day 64 (only for multiple high repeat dose group).
  Incidence and severity of local reactions (pain, tenderness, erythema, swelling, other e.g., ulceration, scabs, bruising, itching and paraesthesia) at the site of vaccination; Incidence and severity of systemic reactions (fatigue, myalgia, malaise, fever, rigors, arthralgia, nausea, diarrhea, light-headedness, dizziness, hypersensitivity and headache). Any 'solicited' AE with onset outside the specified 7-day period of follow-up will be reported as an unsolicited AE.
Occurrence of AEs | From baseline (Day 1) to the end of the 7-day, 28-day follow up period after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment.
Occurrence of any AE during a 60-minute post-vaccination safety observation period | On Day 1 (all cohorts), Day 29 (all cohorts) and Day 57 (Cohort 3 only)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment.
Occurrence of any AE leading to withdrawal | During the 28-day follow up period after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment.
Occurrence of any serious adverse event (SAE) | From baseline (Day 1) to the last visit, assessed up to 14 months
  A SAE is any untoward medical occurrence that, at any dose: • Results in death; • Is life-threatening, (NOTE: The term 'life-threatening' in the definition of 'serious' refers to an event/reaction in which the participant was at risk of death at the time of the event/reaction; it does not refer to an event/reaction which hypothetically might have caused death, if it were more severe); • Requires inpatient hospitalization or prolongation of an existing hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Is a medically important event or reaction.
Occurrence of any clinically significant clinical laboratory abnormalities | From baseline (Day 1) to the last visit, assessed up to 14 months
  Measured as Toxicity Grade ≥1.
Treatment-emergent, clinically significant changes in vital signs and physical examinations. | At specified intervals after each vaccination on Day 1 (all cohorts), Day 29 (all cohorts) and Day 57 (Cohort 3 only)
  Vital signs include systolic and diastolic blood pressures, respiratory rate, pulse rate and oral temperature.

SECONDARY OUTCOMES:
Humoral response to BARS13 | Prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only)
  IgG antibody titres measured by enzyme-linked immunosorbent assay (ELISA) prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only), as well as at follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose, expressed as follows: Corrected post-dose GMTs of IgG (GP)
Humoral response to BARS13 | At follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose
  IgG antibody titres measured by enzyme-linked immunosorbent assay (ELISA) prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only), as well as at follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose, expressed as follows: Corrected post-dose GMTs of IgG (GP)
Humoral response to BARS13 | Prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only)
  IgG antibody titres measured by enzyme-linked immunosorbent assay (ELISA) prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only), as well as at follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose, expressed as follows: Post-dose geometric mean fold rises (GMFRs) from baseline of IgG (GP)
Humoral response to BARS13 | At follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose
  IgG antibody titres measured by enzyme-linked immunosorbent assay (ELISA) prior to each vaccination (Day 1 and Day 29 for all cohorts, and Day 57 for Cohort 3 only), as well as at follow-up visits at 4, 8, 16, 24, 32, 40 and 52 weeks post last dose, expressed as follows: Post-dose geometric mean fold rises (GMFRs) from baseline of IgG (GP)

OTHER OUTCOMES:
Blood samples for exploratory immunological analyses | On Day 1 (all cohorts), Day 29 (all cohorts) and Day 57 (Cohort 3 only)
  Blood samples will be collected at time points described in the study schedule for exploratory immunological analyses of the humoral response and CMI to BARS13 by measuring: RSV neutralization activity
Blood samples for exploratory immunological analyses | On Day 1 (all cohorts), Day 29 (all cohorts) and Day 57 (Cohort 3 only)
  Blood samples will be collected at time points described in the study schedule for exploratory immunological analyses of the humoral response and CMI to BARS13 by measuring: CMI PBMC analysis
Blood samples for exploratory immunological analyses | In participants presenting with symptoms to the general practitioner from baseline (Day 1) to the last visit, assessed up to 14 months
  Blood samples will be collected at time points described in the study schedule for exploratory immunological analyses of the humoral response and CMI to BARS13 by measuring: Percentage of participants with RSV-mediated infection detected by: RT-PCR
Blood samples for exploratory immunological analyses | At follow-up visits 4, 8, 16, 24, 32, 40 and 52 weeks post last dose
  Blood samples will be collected at time points described in the study schedule for exploratory immunological analyses of the humoral response and CMI to BARS13 by measuring: Percentage of participants with RSV-mediated infection detected by: IgM (NP)
Blood samples for exploratory immunological analyses | At follow-up visits 4, 8, 16, 24, 32, 40 and 52 weeks post last dose
  Blood samples will be collected at time points described in the study schedule for exploratory immunological analyses of the humoral response and CMI to BARS13 by measuring: Percentage of participants with RSV-mediated infection detected by: IgG (NP)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Martin, MBBS, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd, Herston, Queensland
  - CMAX Clinical Research, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No
The results of this clinical trial may be published or presented at scientific meetings. If this is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. The Sponsor will comply with the requirements for publication of clinical trial results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicentre studies only in their entirety and not as individual site data. In this case, a coordinating Investigator will be designated by mutual agreement. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.